CLINICAL TRIAL: NCT05396495
Title: Safety and Initial Feasibility of Using the Neurolyser XR Device for the Treatment of Sacroiliac Joint Related Low Back Pain
Brief Title: Safety and Feasibility of the NeurolyserXR for Sacroiliac Joint Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FUSMobile Inc. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIJ-001
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Sacroiliitis
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Intervention Model Description: Pilot, Interventional, Prospective, Open label, Single Arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Treatment arm using the NeurolyserXR to non-invasively ablate the posterior sacral branches enervating the sacroiliac joint
  Interventions: Device: NeurolyserXR

INTERVENTIONS:
Device: NeurolyserXR — Using the NeurolyserXR to non-invasively ablate the posterior sacral branches enervating the sacroiliac joint

SUMMARY:
Pilot study to evaluate the safety and the effectiveness of the Neurolyser XR as a treatment for sacroiliitis

DETAILED DESCRIPTION:
Pilot, Interventional, Prospective, Open label, Single Arm study to evaluate Non-invasive thermal ablation of the posterior sacral nerve branches as a treatment of painful sacroiliac joint (SIJ) using High Intensity Focused Ultrasound delivered by the Neurolyser XR.

Patient would be treated and then followed for up to 6 months. Primary safety endpoint will be measured by the incidence and severity of treatment related adverse events Primary effectiveness endpoint will be measured by the changes in average pain score and Rolland Morris Disability Questionnaire between baseline and 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and females, legally able and willing to participate in the study and come for follow-up visits
2. Able and willing to fill the research questionnaires and to communicate with investigator and research team
3. Patient with bilateral or unilateral sacroiliac joint pain of > 6 months duration
4. Patients presenting with a) a positive (>70% pain relief) to a previous nerve ablation procedure of the sacroiliac joint and / or b) with a positive (>70% pain relief) to a previous nerve block procedure of the sacroiliac joint within the last six months)
5. Average pain score of 4 or higher in the last month, (on 0-10 scale).

Exclusion Criteria:

1. Pregnant or breastfeeding patient
2. Patients younger than 18 or older than 80 years
3. Patients presenting with neurological deficits (including lumbosacral radiculopathy but not solitary radicular pain).
4. Patients with history of lumbar and / or sacral spine surgery
5. Patients with the presence of metal hardware at the lumbosacral spine
6. Patients with history of pelvic pathology that may increase procedural risk and / or influence symptoms and / or generate unrelated adverse event (per the discretion of the study PI)
7. Patients unable to understand and complete the research questionnaires in Hebrew.
8. Patients presenting with any severe medical condition preventing the patient from safely and effectively being treated in the study or reporting study outcome.
9. Patient with extensive scarring in the skin and tissue overlying the treatment area.
10. Patients enrolled in or planned to be enrolled in another clinical trial during the duration of this research project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness per pain score using numerical rating scale of 0 to 10 | Baseline throughout the follow-up period of six months
  Pain reduction would be measured using numerical rating scale of 0 to 10 to evaluate pain and brief pain inventory questioner
Safety per adverse events | Baseline throughout the follow-up period of six months
  Measured by the incidence and severity of treatment related adverse events

SECONDARY OUTCOMES:
Assess self-rated physical disability caused by low back pain | Baseline throughout the follow-up period of six months
  Roland-Morris Disability Questionnaire providing a scale of 0 to 24 when 0 is best and 24 is worst
Opioid intake dosage using morphine equivalency conversion | Baseline throughout the follow-up period of six months
  Using by recording patient opioid intake using opioid equivalency chart

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Giv‘atayim, Israel

IPD SHARING:
Plan to Share IPD: No